CLINICAL TRIAL: NCT02144194
Title: TNM Trial: Upfront Docetaxel [T] and Alternating iv and Oral Vinorelbine [N] Followed, by Either Maintenance Oral Vinorelbine, or Observation for Advanced Breast Cancer
Brief Title: Maintenance Oral Vinorelbine or Observation After Vinorelbine-Docetaxel First Line Chemotherapy in Advanced Breast Ca
Acronym: TNM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Research Group - Collaborative Group, Beirut, Lebanon. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRG SE036
Record Dates: First submitted 2014-05-15; First posted 2014-05-21 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: Oral Vinorelbine; Oral Chemotherapy; Metastatic Breast Cancer; Advanced Breast Cancer; Maintenance treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maintenance treatment (Experimental): Initial treatment Vinorelbine-Docetaxel Vinorelbine I.V: 20mg/m2 D1 Docetaxel: 60mg/m2 D1 Vinorelbine Oral: 60mg/m2 D8 Every 3 weeks for 6 cycles
  Followed by:
  Oral Vinorelbine 60mg/m2 D1, D8 or 80mg/m2 D1, D8 (dose schedule at investigator's discretion) Every 3 weeks until disease progression, unacceptable toxicities or patient refusal to continue
  Interventions: Drug: Vinorelbine-Docetaxel; Drug: Vinorelbine
- Observation arm (Experimental): Initial treatment: Vinorelbine-Docetaxel Vinorelbine I.V: 20mg/m2 D1 Docetaxel: 60mg/m2 D1 Vinorelbine Oral: 60mg/m2 D8 Every 3 weeks for 6 cycles
  Patients in the observation arm will not be administered any treatment after Vinorelbine-Docetaxel
  Interventions: Drug: Vinorelbine-Docetaxel

INTERVENTIONS:
Drug: Vinorelbine-Docetaxel — Vinorelbine I.V: 20mg/m2 D1 Docetaxel: 60mg/m2 D1 Vinorelbine Oral: 60mg/m2 D8 Every 3 weeks x 6 cycles
  Other Names: Navelbine; Navelbine IV; Navelbine Oral; Taxotere
Drug: Vinorelbine — Oral Vinorelbine 60mg/m2 or 80mg/m2 D1, D8 every 3 weeks until disease progression, unacceptable toxicities or patient refusal to continue (dose schedule is at investigator's discretion)
  Other Names: Navelbine Oral
  Arms: Maintenance treatment

SUMMARY:
This 2 arms study will assess the efficacy and safety of the Vinorelbine-Docetaxel combination given as an initial upfront treatment (first line) to all metastatic breast cancer patients enrolled. Patients having a disease control following initial treatment, will be randomized to either oral Vinorelbine maintenance arm or Observation arm. The trial will also compare the efficacy and safety of maintenance oral Vinorelbine versus Observation.

DETAILED DESCRIPTION:
To our knowledge, this is the first trial evaluating the role of oral Vinorelbine as a maintenance therapy versus observation following a first line treatment with iv/oral Vinorelbine+Docetaxel. Eligible patients will be enrolled in the trial to receive 6 cycles of iv(D1)/oral(D8) Vinorelbine + Docetaxel. For responding and SD patients, after the 6 cycles, they will be randomized either in observation arm or to receive a maintenance chemotherapy with oral Vinorelbine. The oral form of the drug was found to be most appropriate for a long term treatment allowing to preserve QoL of the patients. Oral Vinorelbine will be administered on D1, D8 every 3 weeks during maintenance treatment, until PD, unacceptable toxicity or patient refusal to continue. The trial will assess efficacy/safety of initial Vinorelbine-Docetaxel combination as well as the benefits of maintenance chemotherapy with oral Vinorelbine.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients >=18 years of age
* Histologically or cytologically confirmed adenocarcinoma of the breast that is now metastatic or locally-recurrent and inoperable with curative intent
* Measurable and/or non-measurable disease
* The patient's primary and/or metastatic tumor is HER2 neu negative
* Documented metastatic disease previously untreated with palliative chemotherapy
* Adjuvant or neo-adjuvant chemotherapy (including treatment with docetaxel or any other chemotherapy) is allowed with a disease free survival of at least 6 months
* No symptom or sign of brain metastasis

Exclusion Criteria:

* Operable local recurrence
* Ascites or pericardial effusion as only site of metastasis
* Symptomatic peripheral neuropathy > grade 1 according to the NCI Common Toxicity Criteria
* Radiotherapy to all areas of evaluable disease within the previous 4 weeks
* Disease significantly affecting absorption
* Severe hepatic insufficiency
* Patient previously treated with chemotherapy for their metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Time To Disease Progression of patients who are treated with Vinorelbine-Docetaxel followed by maintenance oral Vinorelbine vs patients treated with Vinorelbine-Docetaxel without maintenance treatment | Up to 36 months

SECONDARY OUTCOMES:
Overall Response Rate | Up to 36 months
Duration of Response | Up to 36 months
Quality of Life | Up to 36 months
Number and percentage of participants with Adverse Events | Participants will be followed for the entired duration of the study, an expected average of 60 months
3-Y Overall Survival | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Fadi Farhat, M.D, Principal Investigator — Hammoud Hospital University Medical Center; Marwan Ghosn, M.D, Principal Investigator — Hotel Dieu De France University Hospital; Georges Chahine, M.D, Principal Investigator — Hotel Dieu de France University Hospital; Joseph Kattan, M.D, Principal Investigator — Hotel Dieu de France University Hospital; Nizar Bitar, M.D, Principal Investigator — Sahel General Hospital
Locations (2):
- Lebanon (2):
  - Hotel Dieu de France University Hospital, El Achrafiyé, Beyrouth
  - Hammoud Hospital University Medical Center, Saida, Saida

IPD SHARING:
Plan to Share IPD: No